CLINICAL TRIAL: NCT07238725
Title: The Efficacy of Aldehyde Dehydrogenase Enzyme in Essential Tremor Patients: A Single-Center Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Pico Entech Co., Ltd. (Industry)
Collaborators: Korea University Anam Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024AN0506; NCT07124507 (obsolete NCT alias)
Record Dates: First submitted 2025-10-23; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Essential Tremor
Keywords: Essential Tremor; Tremor; ALDH; Aldehyde Dehydrogenase; Oxidative Stress; Antioxidant
MeSH Terms: conditions — Essential Tremor; Tremor

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label trial
Masking Description: Open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALDH Food Supplement (Experimental): Participants in this arm will receive an ALDH-containing food supplement (PICOZYME ET) twice daily for 3 months. The study will assess changes in tremor severity, quality of life, and exploratory metabolic biomarkers.
  Interventions: Dietary Supplement: PICOZYME ET

INTERVENTIONS:
Dietary Supplement: PICOZYME ET — The investigational product is a dietary supplement containing aldehyde dehydrogenase (ALDH), administered orally twice daily (one packet in the morning and one in the evening) for 3 months before meals.
  Other Names: ALDH food supplement

SUMMARY:
This is a sponsor-initiated, single-arm, single-center clinical trial designed to evaluate the efficacy and safety of an ALDH-containing food supplement (PICOZYME ET) in patients with Essential Tremor (ET). Participants will consume the investigational product daily for three months, and clinical outcomes will be assessed using the Clinical Rating Scale for Tremor (CRST) and the Activities of Daily Living (ADL) scale. Additional exploratory analyses will evaluate changes in metabolic biomarkers and brain function via imaging and blood tests.

DETAILED DESCRIPTION:
Essential Tremor (ET) is one of the most common adult movement disorders, characterized by involuntary rhythmic tremors, primarily affecting the hands. Although not life-threatening, ET significantly impacts quality of life and daily functioning. Recent studies suggest that oxidative stress and impaired GABAergic inhibition may be involved in its pathophysiology, and aldehyde dehydrogenase (ALDH) is believed to play a role in mitigating these mechanisms.

This single-center, open-label, sponsor-initiated study is funded by PICO Entech Corp and conducted at Korea University Anam Hospital under the supervision of the institutional IRB. The trial aims to evaluate the efficacy and safety of an ALDH-containing food supplement (PICOZYME ET) in patients with ET. A total of 40 adult participants diagnosed with ET will be enrolled and instructed to consume the investigational food product twice daily for three months. Efficacy will be measured by changes from baseline in the Clinical Rating Scale for Tremor (CRST) and Activities of Daily Living (ADL) scores.

Secondary outcomes include safety and biomarker analysis through blood tests. Exploratory outcomes include changes in metabolic activity via FDG PET-CT imaging, levels of oxidative stress biomarkers (malondialdehyde, total aldehyde), and potential associations with GABA-related metabolic pathways.

The study has received IRB approval from Korea University Anam Hospital and includes oversight from a Data Safety Monitoring Board (DSMB). All participants will provide written informed consent before enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 19 years who provide written informed consent.
* Diagnosed with Essential Tremor (ET) by a board-certified neurologist or neurosurgeon.
* Presence of postural or intention tremor in the dominant hand/arm with a CRST score ≥ 2.
* Stable medication regimen for at least 30 days prior to enrollment.
* No structural brain abnormalities on MRI within the last 3 years.
* Eligible according to investigator assessment and agreement by two clinical team members.

Exclusion Criteria:

* Presence of secondary tremor causes (e.g., Parkinsonism, dystonia).
* Significant medical conditions such as severe arrhythmia, renal failure, hepatic failure, acute stroke, or epilepsy.
* Contraindications to MRI (e.g., pacemakers, metal implants).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Rating Scale for Tremor (CRST) total score from baseline to 3 months | Baseline and 3 months
  The CRST is a validated clinical tool used to quantify tremor severity. It includes assessments of postural, action, and intention tremor, as well as functional disability. Total scores range from 0 to 160, with higher scores indicating more severe tremor.
Change in Activities of Daily Living (ADL) score from baseline to 3 months | Baseline and 3 months
  ADL will be assessed using the QUEST (Quality of Life in Essential Tremor) questionnaire. Higher scores indicate greater functional impairment.

SECONDARY OUTCOMES:
Change in 24-hour Urinary Catecholamine Levels (epinephrine, norepinephrine, dopamine) | Baseline and 3 months
  Measurement of 24-hour urinary catecholamine levels (epinephrine, norepinephrine, dopamine) in µg/day at baseline and 3 months to evaluate oxidative stress.
Change in Random Urinary Malondialdehyde | Baseline and 3 months
  Semi-quantitative measurement of malondialdehyde in random urine using dipstick analysis (DFI FRC 50SF analyzer and Free RadiCheck test strips), with results reported as relative values.
Change in Serum C-Reactive Protein (CRP) Level | Baseline and 3 months
  Measurement of serum CRP concentration in mg/L at baseline and 3 months.
Incidence of adverse events during the intervention period | Through study completion (up to 3 months)
  Adverse events (e.g., nausea, gastrointestinal discomfort) will be monitored and recorded throughout the 3-month supplementation period to assess safety.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. This study involves a small, single-site intervention, and data sharing is not planned due to institutional policy and privacy considerations.

REFERENCES:
- [Result] Louis ED, Ferreira JJ. How common is the most common adult movement disorder? Update on the worldwide prevalence of essential tremor. Mov Disord. 2010 Apr 15;25(5):534-41. doi: 10.1002/mds.22838. PMID 20175185
- See also: Related Info — https://picoentech.com/